CLINICAL TRIAL: NCT02345239
Title: Impact of Pantoprazole on 24-H Glycemic Control and on Post-prandial Glucose Excursion Inpatients With Type 2 Diabetes
Brief Title: Impact of Pantoprazole on 24-H Glycemic Control and on Post-prandial Glucose Excursion in Patients With Type 2 Diabetes
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr. Waheed Rehman (Other)
Responsible Party: Sponsor-Investigator, Dr. Waheed Rehman, Physician/Resident, McGill University
Organization: McGill University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-329-BMB
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Pantoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pantoprazole (Experimental): Pantoprazole
  Interventions: Drug: Pantoprazole

INTERVENTIONS:
Drug: Pantoprazole — proton pump inhibitor

SUMMARY:
The purpose of this study is to demonstrate the immediate impact of pantoprazole on 24-H glycemic control and on post-prandial glucose excursion in patients with type 2 diabetes.If our data support the previous animal, observational and clinical studies results, PPIs could become a new anti-diabetic agent with a good and safe profile for type 2 diabetes

DETAILED DESCRIPTION:
Diabetes mellitus is a complex chronic disease associated with an absolute insulin deficiency in type1 diabetes and a progressive deterioration of b-cell function in type 2 diabetes. The pathophysiology of type 2 diabetes includes not only the classical insulin resistance in muscle and liver and progressive b-cell failure but also accelerated lipolysis, incretin deficiency/resistance, hyperglucagonemia, renal increased glucose reabsorption, and brain insulin resistance. Finally, hyperglycemia in both type 1 and 2 diabetes results from an absolute or relative deficit in the pancreatic b -cell mass.

Gastrin has long been considered a candidate incretin hormone, i.e. an enteral factor responsible for the more than 2-fold increase in insulin secretion when glucose is ingested orally than when administered intravenously to match peripheral glucose levels. In healthy humans, acute administration of gastrin to achieve supraphysiological levels leads to a modest release of insulin under basal glucose conditions and a more pronounced potentiation of insulin release when coadministered with glucose. With the identification of gastric inhibitory polypeptide, now known as glucose-dependent insulinotropic polypeptide, and subsequently glucagon-like peptide-1 as more potent incretin hormones whose secretion may be impaired in type 2 diabetes, attention largely shifted away from gastrin playing an important role in the enteroinsular axis.

Like gastric inhibitory polypeptide and glucagon-like peptide-1, gastrin has also been shown to induce b-cell proliferation and neogenesis in various model systems, and also appears to increase the insulin content of individual cells. Zollinger and Ellison's original description of peptic ulcer disease attributable to purported gastrinoma included one case where "the pancreatic tissue removed with the tumor showed normal islands with many large cells…". Examination of another case with resected pancreas adjacent to an antral gastrinoma "showed a marked proliferation of ducts and islet tissue" with "development of islets from cells (nesidioblasts) within the duct epithelium.

Gastrin has demonstrated to be an islet growth factor (like glucagon-like peptide, epidermal growth factor, transforming growth factor) and be able to restore a functional b-cell mass in diabetic animals.

This combination drug therapy, specifically sitagliptin and pantoprazole, induces b-cell neogenesis in adult human pancreatic cells implanted in NOD-severe combined immunodeficient mice. The increased b-cell mass appears to be derived from pancreatic exocrine duct cells.

PPIs have also demonstrated a positive effect on glycemic control in a model of type 2 diabetes-Psammomys obesus. In this study PPI lansoprazole had significant glucose-lowering effects in an animal model of type 2 diabetes, an effect that is most likely mediated through an increase in endogenous gastrin levels.

In summary basic research demonstrated that gastrin can be considered as an important regulator of b-cell neogenesis and glucose homeostasis. Neogenesis by the process of transdifferentiation appears to be activated only after severe injury to endocrine or exocrine pancreatic tissue, or when strong additional stimuli like GLP-1 and/or gastrin are provided.

All the retrospective studies showed antidiabetic properties for the PPIs with a global glucose-lowering power around 0.6-0.7 % points of HbA1c, but the level of evidence for the available literature is still not high.

Moreover, studies in endogenous hypergastrinemia support an incretin effect of gastrin in man. All the basic research shows gastrin has a significant role in BG control by Beta cell proliferation, increase insulin secretion particularly post prandial peak and incretin like action. The findings of this study provide modest support for the proposition that PPIs may be a useful adjunctive therapy for type 2 diabetes. The postulated mechanism for this effect is PPI causing elevation of serum gastrin, enhancing pancreatic β-cell function, and stimulating increased insulin secretion. Proton pump inhibitors (PPIs) can raise serum gastrin concentration significantly and therefore, affect to glucose metabolism through promoting b-cell regeneration/expansion and also enhancing insulin secretion.

The results of different observational studies showed anti-diabetic properties for the PPIs with a global glucose-lowering power around 0.6-0.7 % points of HbA1c. Small clinical trials have proved that PPI have significant impact on fasting blood glucose, HbA1C, C-peptides and beta cell mass. In most of the trials there was significant drop in fasting blood glucose after 12 weeks of PPI but post prandial and immediate effects were not explored.

The purpose of this study is to demonstrate the immediate impact of pantoprazole on 24-H glycemic control and on post-prandial glucose excursion in patients with type 2 diabetes. This study can be extended to 12 weeks period and see the long term impact of PPI on post prandial glucose and HbA1C. If our data support the previous animal, observational and clinical studies results, PPIs could become a new anti-diabetic agent with a good and safe profile for type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria: Type 2 Diabetes with HbA1C > 8% -

Exclusion Criteria: Type diabetics 1 and 2 on insulin

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Mean 24-hour glucose level | 7 days
Mean post-prandial glucose excursion | 7 days

SECONDARY OUTCOMES:
Mean Mean 24-hour glucose level | day 6 and 7
  after discontinuation of pantoprazole
Postprandial glucose excursion | day 6 and 7
  after discontinuation of pantoprazole

CONTACTS AND LOCATIONS:
Overall Officials: Waheed Rehman, FRCPC,DABIM, Principal Investigator — McGill University

REFERENCES:
- [Background] Defronzo RA. Banting Lecture. From the triumvirate to the ominous octet: a new paradigm for the treatment of type 2 diabetes mellitus. Diabetes. 2009 Apr;58(4):773-95. doi: 10.2337/db09-9028. No abstract available. PMID 19336687
- [Background] Allen JM, Adrian TE, Webster J, Howe A, Bloom SR. Effect of single dose of omeprazole on the gastrointestinal peptide response to food. Hepatogastroenterology. 1984 Feb;31(1):44-6. PMID 6365714
- [Background] Bellomo Damato A, Stefanelli G, Laviola L, Giorgino R, Giorgino F. Nateglinide provides tighter glycaemic control than glyburide in patients with Type 2 diabetes with prevalent postprandial hyperglycaemia. Diabet Med. 2011 May;28(5):560-6. doi: 10.1111/j.1464-5491.2010.03219.x. PMID 21204958
- [Background] Bodvarsdottir TB, Hove KD, Gotfredsen CF, Pridal L, Vaag A, Karlsen AE, Petersen JS. Treatment with a proton pump inhibitor improves glycaemic control in Psammomys obesus, a model of type 2 diabetes. Diabetologia. 2010 Oct;53(10):2220-3. doi: 10.1007/s00125-010-1825-6. Epub 2010 Jun 30. PMID 20585936
- [Background] Boj-Carceller D. Proton pump inhibitors: impact on glucose metabolism. Endocrine. 2013 Feb;43(1):22-32. doi: 10.1007/s12020-012-9755-3. Epub 2012 Aug 12. PMID 22886351
- [Background] Boj-Carceller D, Bocos-Terraz P, Moreno-Vernis M, Sanz-Paris A, Trincado-Aznar P, Albero-Gamboa R. Are proton pump inhibitors a new antidiabetic drug? A cross sectional study. World J Diabetes. 2011 Dec 15;2(12):217-20. doi: 10.4239/wjd.v2.i12.217. PMID 22174957
- [Background] Brand SJ, Tagerud S, Lambert P, Magil SG, Tatarkiewicz K, Doiron K, Yan Y. Pharmacological treatment of chronic diabetes by stimulating pancreatic beta-cell regeneration with systemic co-administration of EGF and gastrin. Pharmacol Toxicol. 2002 Dec;91(6):414-20. doi: 10.1034/j.1600-0773.2002.910621.x. PMID 12688387
- [Background] Brunner G, Athmann C, Schneider A. Long-term, open-label trial: safety and efficacy of continuous maintenance treatment with pantoprazole for up to 15 years in severe acid-peptic disease. Aliment Pharmacol Ther. 2012 Jul;36(1):37-47. doi: 10.1111/j.1365-2036.2012.05106.x. Epub 2012 Apr 24. PMID 22531114
- [Background] Crouch MA, Mefford IN, Wade EU. Proton pump inhibitor therapy associated with lower glycosylated hemoglobin levels in type 2 diabetes. J Am Board Fam Med. 2012 Jan-Feb;25(1):50-4. doi: 10.3122/jabfm.2012.01.100161. PMID 22218624